CLINICAL TRIAL: NCT01225497
Title: Effects of Two Eccentric Exercise Protocols on Reported Pain Intensity, Function, and Treatment Satisfaction in Adults With Chronic Mid-portion Achilles Tendinopathies
Brief Title: Eccentric Exercise for Chronic Mid-portion Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Margaret University (Other)
Responsible Party: Mr Marc Stevens/Highly Specialist Physiotherapist, NHS Forth Valley / Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FV526
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: Achilles Tendon; Tendinopathy
Keywords: Randomized; Pilot study; VISA-A; VAS
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard eccentric exercise (Active Comparator): Participants randomised to this group shall complete 180 repetitions a day of Alfredsons heel drop protocol. This has been accepted as standard management for mid-portion Achilles pain in the first instance.
  Interventions: Procedure: Standard eccentric exercise
- Eccentric exercise as able (Experimental): Participants randomised to this group shall carry out exactly the same eccentric exercises as per Alfredsons heel drop protocol. However, these individuals will be instructed to do what they can.
  Interventions: Procedure: Eccentric exercise-Experimental group

INTERVENTIONS:
Procedure: Standard eccentric exercise — Participants stand with the balls of their feet on a step. They rise up onto tip toes using both legs then transfer onto the affected leg, then slowly lower their heel below the level of the step keeping their weight-bearing limb fully straight (eccentric phase). This constitutes 1 repetition and is repeated for 3 x 15 reps.
  The previous procedure is then carried out with the knee bent during the eccentric phase of loading for 3 x 15 reps.
  All of the above is carried out twice a day as per Alfredsons protocol. Participants are encouraged as per Alfredsons procedure to continue into discomfort not severe pain.
  Arms: Standard eccentric exercise
Procedure: Eccentric exercise-Experimental group — Eccentric exercise is performed the same as in the standard group. However participants in this group are encouraged to do the number of repetition they can manage so long as it is also to discomfort.
  Arms: Eccentric exercise as able

SUMMARY:
Chronic pain and disability are unfortunately common in Achilles tendon pain. Outcome after surgery is often poor. Also tendon pain can be resistant to treatment and may lead to cessation of hobbies or careers.

Recently eccentric exercise (defined as muscle loading where tension develops as physical lengthening occurs) has become a cornerstone in managing tendon pain due to an increasing amount of favorable research. Eccentric exercises are considered to be non-invasive, safe, and appear to be important for a successful outcome.

One exercise program has been extensively adopted in research and clinical practice for Achilles pain. It recommends individuals perform 180 repetitions a day. However there appears to be little scientific rationale for this number. Consequently there may be significant implications for patient compliance, satisfaction, and overall treatment efficacy in a strategy which is encouraged to be uncomfortable.

Fifty two adults (18-70 years old), with mid-Achilles tendon pain will be randomised to standard treatment (180 repetitions) or to a group where individuals are allowed to do what they can. Participants will be recruited from participating physiotherapy departments (health centres and hospital departments) across NHS Forth Valley. All individuals will be required to complete the same type of eccentric exercise for six weeks attending an initial assessment and two follow-up appointments at three and six weeks. Thereafter participants will be discharged if better, or continue with individual care where appropriate.

It is hoped this pilot study will establish if future larger scale investigation is warranted examining whether it is necessary to subject individuals to 180 repetitions a day in an activity recommended to be uncomfortable. Also will participant satisfaction differ between exercise groups? If further investigation is warranted this pilot may provide population specific data for future sample size calculations, and may provide a suitable methodology for such investigations.

DETAILED DESCRIPTION:
Design: This project will be a prospective double-blinded randomised clinical controlled trial comparing a "standard" volume eccentric exercise program (Group I-Control) versus a participant determined volume program (Group II-Experimental).

Participants Participant population The participant population of interest are those attending NHS out-patient physiotherapy departments for the treatment of chronic mid-portion Achilles tendinopathy in Scotland. Consequently both genders and varying pre-morbid activity levels will be anticipated across a wide age range.

Participant recruitment and selection Physiotherapy colleagues across Forth Valley NHS Trust will be contacted via a standardised email inviting individuals to participate in the proposed investigation. Those volunteering will be required to identify potential participants currently waiting to attend physiotherapy. Such waiting lists include self-referral, orthopaedic and GP referrals.

Once identified potential participants will be sent standardised letters of introduction identifying they may be eligible to participate in a research project concerning physiotherapy treatment of Achilles tendon pain. More detailed participant information sheets will also be included to allow candidates have best opportunity to provide informed consent. Any potential risks will be outlined. As part of the informed consent process participants will be encouraged to seek opinions from friends and family. Participant recruitment will be implemented over a 4 month period. Potential participants will be instructed that they will receive an appointment in due course at the location they would normally attend.

On initial contact participants will be assessed as per normal practice by participating physiotherapists in the health centres or hospitals they would normally attend in an attempt to minimise disruption to the patient journey. It is hoped travel will be minimised for participants in order to minimise drop out and participant expense. In instances where diagnosis is uncertain participating therapists are advised to seek a second opinion from appropriate colleagues/senior clinical staff as they would do under normal circumstances. If a diagnosis of Achilles tendinopathy is still uncertain the potential participant will not be included and will be informed why. Participating therapists will undergo training in obtaining informed consent; diagnosing Achilles tendinopathy as defined in the following inclusion criteria; and receive instruction in data collection procedures required for this investigation from the principle researcher.

Again any potential risks will be outlined in the process of obtaining informed consent. Participants will be given time to consider their options. It will be made clear that deciding not to participate will not affect future treatment. If potential participants agree to take part, eligibility to participate will be assessed against the following criteria. If potential participants are suitable they will then be randomised to either group. Participants will be reminded of their right to withdraw from the trial at anytime and this will not affect future treatment. If necessary on withdrawal participants will be informed that they can request to be seen by a different physiotherapist if they so wish. If an individual does not fulfil the selection criteria they will be informed why immediately and then managed as per normal.

Sampling technique It is anticipated the sample size required will be obtained. Nevertheless, due to uncertain incidence rates and the limited time convenience sampling will be used to maximise recruitment.

Participant randomisation Once recruited, participants will be randomised to the control group ("standard" volume) or experimental group (patient determined volume). Randomisation will be achieved by participating physiotherapists telephoning a recruited Stirling Royal Infirmary physiotherapy department secretary at the end of the initial consultation. The secretary will randomly draw sealed opaque envelopes detailing the number of repetitions to do per day and inform the participant directly. As well as written documentation provided at the initial consultation the participant will be reminded not to discuss the volume of repetitions with anyone potentially participating in the trial or with the participating therapist for the duration of testing. In this way the participants, participating therapists and researcher will be blinded to group allocation. Any questions participants may have will be directed to the independent supervisor of the project (Frank Gilroy, Physiotherapy Manager, Forth Valley NHS Trust).

Sample size calculation The VISA-A has been suggested to be valid and reliable and is therefore strongly recommended for use when researching and treating Achilles tendon pain (Robinson 2001; Brukner & Khan 2007). Thus it will be used as the principle outcome measure of this investigation. Previous research suggests a delta of 10 points with a standard deviation of 12 when comparing eccentric exercise to a wait and see approach (Rompe et al 2008) giving a large effect size of 0.83. With a power of 0.80, an alpha level of 0.05, and using methods outlined by Fleiss (1986) it is calculated that 23 participants are required for each group of this trial. All studies in this area assign an additional 10% to the calculated sample size to account for loss to follow-up (Rompe et al 2007). This appears to be adequate for the proposed population and setting as no studies have failed to recruit the required number to ensure adequate power. Therefore a total of 26 patients will be required for each arm of this trial.

Procedure Participants will be assessed, recruited and randomised as detailed previously. All participants will be instructed in the same eccentric exercise technique as per previous literature (Alfredson et al 1998). Advice concerning progression, and exercising to pain will be consistent across groups with that recommended by Alfredson et al (1998). All participants will also receive the same written instructions on how to perform and progress exercise as well as a simple exercise diary to record the number of repetitions actually completed per day. During the initial consultation the data collection sheet will be completed where appropriate. At the end of the initial consultation participating therapists will phone Stirling Royal Infirmary physiotherapy department where the recruited secretary will inform the patient directly the number of exercises to do a day (as part of the randomisation process). A follow-up appointment will be arranged in three weeks.

At week three exercises will be reviewed to ensure good technique. All outcome measures will be re-assessed and documented on the data collection sheet.

At week six all outcome measures will be re-assessed. Patient satisfaction with treatment will be assessed. All completed data collection sheets and exercise activity logs will be mailed to the principle investigator for analysis. At this point participants will be informed the trial is over and management will continue as per normal practice. If symptoms have resolved participants may be discharged; if they are improving they may be given an open appointment with advice to contact if any further problems; if there is little change therapists will be allowed to continue management as they see fit as per normal practice.

At the end of the trial the principle researcher will attempt to contact participants lost to follow-up to determine any reasons for this as long as they have agreed to this during the consenting process.

ELIGIBILITY:
Inclusion Criteria:

* Mid-portion Achilles tenderness on palpation or during/after activity 2-7cm proximal to insertion of a month or more duration
* Wish to return to previous level of function
* Tendon thickening 2-7cm proximal to insertion may or may not be present. Although associated with Achilles tendinopathies it is not required for diagnosis
* 18-70 years of age
* Ability to give informed written consent

Exclusion Criteria:

* Indeterminate diagnosis
* Tendon insertion pain
* Recent fracture of the affected lower limb (within the last 12 months)
* Presence of bursitis
* Less than one month of symptoms
* Previous surgical intervention near the Achilles tendon (within the last 12 months)
* Previous experience of eccentric loading
* Sudden onset of symptoms suggesting partial rupture rather than tendinopathy
* Previous tendon rupture
* Steroid injection near the Achilles tendon in the last month
* Presence of rheumatoid arthritis, diabetes, or other systemic disorders; radiculopathy etc. that could significantly contribute to posterior ankle pain
* Congenital or acquired deformities of the knee or ankle
* Inability to complete eccentric exercises
* Inability to understand spoken or written English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment-Achilles (VISA-A) | Baseline
  The VISA-A is has been reported as a valid and reliable measure for determining the extent of functional limitation in individuals suffering Achilles tendon pain. It has been recommended for use in reseach evaluating Achilles tendon pain. It is a questionnaire which gives a score out of 100 with higher scores indicating increasing levels of disability.
Victorian Institute of Sports Assessment-Achilles (VISA-A) | Week 3
  The VISA-A is has been reported as a valid and reliable measure for determining the extent of functional limitation in individuals suffering Achilles tendon pain. It has been recommended for use in reseach evaluating Achilles tendon pain. It is a questionnaire which gives a score out of 100 with higher scores indicating increasing levels of disability.
Victorian Institute of Sports Assessment-Achilles (VISA-A) | Week 6
  The VISA-A is has been reported as a valid and reliable measure for determining the extent of functional limitation in individuals suffering Achilles tendon pain. It has been recommended for use in reseach evaluating Achilles tendon pain. It is a questionnaire which gives a score out of 100 with higher scores indicating increasing levels of disability.

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline
  This is being utilised in this study to give an indication of the level of intensity of pain an individual with Achilles pain. Participants will make a mark on a 100mm horizontal line to indicate the intensity of their pain.
Participant satisfaction | Week 6
  Simple Likert style descriptors will be used (Poor, moderate, good, excellent).
Visual Analogue Scale | Week 3
  This is being utilised in this study to give an indication of the level of intensity of pain an individual with Achilles pain. Participants will make a mark on a 100mm horizontal line to indicate the intensity of their pain.
Visual Analogue Scale | Weeks 6
  This is being utilised in this study to give an indication of the level of intensity of pain an individual with Achilles pain. Participants will make a mark on a 100mm horizontal line to indicate the intensity of their pain.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Stevens, B.Sc (Hons), Principal Investigator — Queen Margaret University/NHS Forth Valley
Locations (1):
- NHS Forth Valley, Falkirk, United Kingdom

REFERENCES:
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Background] Rompe JD, Furia JP, Maffulli N. Mid-portion Achilles tendinopathy--current options for treatment. Disabil Rehabil. 2008;30(20-22):1666-76. doi: 10.1080/09638280701785825. PMID 18608388
- [Background] Roos EM, Engstrom M, Lagerquist A, Soderberg B. Clinical improvement after 6 weeks of eccentric exercise in patients with mid-portion Achilles tendinopathy -- a randomized trial with 1-year follow-up. Scand J Med Sci Sports. 2004 Oct;14(5):286-95. doi: 10.1111/j.1600-0838.2004.378.x. PMID 15387802
- [Background] Ohberg L, Lorentzon R, Alfredson H. Eccentric training in patients with chronic Achilles tendinosis: normalised tendon structure and decreased thickness at follow up. Br J Sports Med. 2004 Feb;38(1):8-11; discussion 11. doi: 10.1136/bjsm.2001.000284. PMID 14751936